CLINICAL TRIAL: NCT06402162
Title: The Effect of Core Stability Exercises on Pain, Muscle Strength, and Muscle Architecture in Tennis Players With Rotator Cuff Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Emine Merve Ersever, haymana vocational high school physiotherapy, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5678525-050.0404/1202308
Record Dates: First submitted 2024-04-29; First posted 2024-05-07 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-03

CONDITIONS: Exercise; Muscle Weakness; Rotator Cuff Injuries
Keywords: muscle thickness; fiber length; pennation angle; pain
MeSH Terms: conditions — Motor Activity; Muscle Weakness; Rotator Cuff Injuries; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study will include 40 tennis players diagnosed with rotator sheath lesions who meet the inclusion criteria. Groups will be randomly divided into 2. The 1st group will be randomly divided into 2 groups as control (n=20) and 2nd group as core exercise (n=20). Unlike the control group, core exercises will be added to the routine exercise program of tennis players once a day, 3 days a week, for 8 weeks. In both groups, pain will be assessed by Visual Analog Scale (VAS), muscle strength by isokinetic dynamometer and supraspinatus muscle architecture by ultrasonography and dynamic tendon imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- muscle architecture (Experimental)
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — The study will include 40 tennis players diagnosed with rotator cuff lesions who meet the inclusion criteria. The 1st group will be randomly divided into 2 groups as control (n=20) and 2nd group as core exercise (n=20). Unlike the control group, core exercises will be added to the routine exercise program of tennis players once a day, 3 days a week for 8 weeks.

SUMMARY:
This study aims to shed light on the supraspinatus and infraspinatus muscles, which play a significant role in rotator sheath tendinopathy and tears. It includes isometric measurements of muscle thickness, fiber length, and pennation angles, as well as muscle strength, using ultrasound to evaluate the muscle architecture of the supraspinatus and infraspinatus muscles in tennis players.

DETAILED DESCRIPTION:
The shoulder joint is prone to injury due to its unique anatomy. Rotator cuff lesions (RCL) are a common cause of shoulder pain, with a prevalence of 81% (1). One effective approach for monitoring muscle function is to visualize the architectural structure of the muscle. Muscle architecture is the examination of the structural arrangement of muscle fibers, muscle thickness, pennation angle, and number of sarcomeres according to the force generation axis (2). Ultrasonographic muscle architecture measurements provide a rapid and objective evaluation to examine the pathology of the muscles associated with subacromial impingement syndrome (3).

Muscle strength measurement is a physical performance measurement used to determine the loss of strength in the muscle and to evaluate the effectiveness of the intervention by resisting the muscle (4). It is worth noting that the strength of the rotator cuff muscles, especially the external and internal force-generating muscles of the shoulder, may be somewhat reduced in athletes with RCL. Strength measurement of these muscles can provide valuable data in shoulder evaluation (5). It is also worth mentioning that shoulder injuries are quite common in tennis. In addition to physiotherapy methods, the success rate in RCL treatment may be enhanced by exercise (6). In shoulder rehabilitation, core exercises are designed to help restore functional movements through the elimination of pain and the dynamic stability of the rotator cuff and scapular muscles. The goal is to strengthen the shoulder girdle muscles and achieve sufficient joint range of motion, especially by providing neuromuscular re-education with therapeutic exercises.

References

1. Dong W, Goost H, Lin XB, et al. Treatments for shoulder impingement syndrome: a systematic review and network meta-analysis. Medicine (Baltimore). 2015;94:e510.
2. Lewis, J., Ginn, K.. Rotator cuff tendinopathy and subacromial pain syndrome.In: Modern Musculoskeletal Physiotherapy, fourth ed. Elsevier, pp. 2015; 563e568.
3. Michener L, Walsworth M, Burnet E. Effectiveness of rehabilitation for patients with subacromial impingement syndrome: a systematic review. J Hand Ther, 2004, 17: 152-164.
4. Sauers E. Effectiveness of rehabilitation for patients with subacromial impingement syndrome. J Athl Train, 2005, 40: 221-223
5. Ersever, E. M., Güzel, N. A., Hakan, G. E. N. Ç., & Mülkoğlu, C. (2021). Subakromiyal Sikişma Sendromlu Hastalarda Egzersiz İle Elektrik Stimülasyonunun Etkileri. Ankara Eğitim ve Araştırma Hastanesi Tıp Dergisi, 54(3), 382-386.
6. Oh, L.S., Luke, S., Brian, R, Michael P., Bruce, A., Marx, Robert G. (2007). Indications for rotator cuff repair: a systematic review. Clinical Orthopaedics and Related Research®, 455: 52-63.

ELIGIBILITY:
Inclusion Criteria:

* Acute trauma
* Tendinosis
* Bursitis chronic inflammation degeneration
* Grade 1-2 rupture
* Having unilateral shoulder pain
* At least two specific tests must be positive (Neer-hawkings-Lag sign-drop arm and supraspinatus isolation tests; painful shoulder internal and external rotation against resistance (IR and ER); painful arch during abduction)

Exclusion Criteria:

* An acute trauma
* History of surgery or a fracture in or near the shoulder and shoulder
* A neurological deficit
* intra-articular injections in the last six months
* Rheumatic disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
visual pain scale | 8 week
  The primary objective was to see if we could help to decrease the pain intensity of the patients by 4 units in a 10-unit VPS assessment.

SECONDARY OUTCOMES:
ultrasonographic examination | 8 week
  increase in supraspinatus muscle thickness = centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Tennis Club, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Application of core exercises to tennis players — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9740142/pdf/ijerph-19-16033.pdf
- See also: core exercises to tennis players — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9740142/pdf/ijerph-19-16033.pdf